CLINICAL TRIAL: NCT00431756
Title: Novel Biomarkers in the Neoplastic Progression of Barrett's Esophagus (Previously: Methylation in Cancer Progression of Barrett's Esophagus
Brief Title: Novel Biomarkers in the Neoplastic Progression of Barrett's Esophagus
Acronym: BE
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00026956; 1K23DK068149 (NIH)
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Barrett Esophagus; Esophageal Neoplasm; Gastroesophageal Reflux
Keywords: Barrett's esophagus; gastroesophageal reflux disease (GERD); esophageal cancer; DNA methylation
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — approx. 24 ml blood, 1-8 esophageal mucosal pinch specimens and or esophageal brushings
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if there are any early changes in DNA markers of blood and esophageal tissue in people with gastric reflux, Barrett's esophagus or esophageal cancer that can warn of a progression to esophageal cancer.

DETAILED DESCRIPTION:
Patients with Barrett's esophagus (BE) have an increased risk of esophageal adenocarcinoma which is 40-125 fold higher than in the general population. However, the current techniques of detecting dysplasia and observing abnormal p53 immunohistochemical staining are not accurate or reliable methods for determining which BE patients will progress to cancer. DNA hypermethylation is an epigenetic process that occurs in the promoter region of certain genes, resulting in suppression of gene expression. Inactivation of specific genes via hypermethylation has been highly associated with cancer.

The primary objective of this research is to determine whether DNA hypermethylation is a biomarker that will predict which patients with BE are likely to progress to adenocarcinoma. Patients with BE and/or esophageal adenocarcinoma who undergo endoscopy at the Johns Hopkins Hospital will comprise the cohort of subjects. Gene hypermethylation will be assessed by performing methylation-specific Polymerase Chain Reaction (PCR) on a panel of 8 cancer-related genes.

Specific Aim 1: To compare the prevalence of gene hypermethylation in BE patients with different grades of dysplasia and/or adenocarcinoma, using archived specimens.

Specific Aim 2: To determine whether the presence of gene hypermethylation in initial biopsies of BE patients is associated with progression to adenocarcinoma, using archived specimens. To compare gene hypermethylation with currently available markers for neoplastic progression.

Specific Aim 3: To determine whether methylated DNA from BE and/or adenocarcinoma can be detected in the peripheral blood of patients, by comparing methylation profiles of esophageal biopsy specimens with peripheral blood samples taken at the same time in prospectively enrolled patients.

If hypermethylation of one or more genes is detected at an early stage in BE patients who later progress to adenocarcinoma, hypermethylation could be used as an early predictor for adenocarcinoma even before pathologic changes are evident. Furthermore, this research will help determine the specific genetic events that occur in the neoplastic transformation from BE to adenocarcinoma.

The long-term goal of this project is to determine whether hypermethylation can identify BE patients who are at high risk for neoplastic progression, thus allowing for early intervention in the form of more frequent endoscopic surveillance, chemoprevention, ablative therapy, or surgery.

ELIGIBILITY:
Inclusion Criteria:

* People who are undergoing upper endoscopy as part of their medical care with a history of esophageal cancer, Barrett's esophagus, or upper gastrointestinal symptoms.

Exclusion Criteria:

* People who are are currently having chemotherapy, or who have completed chemotherapy within the last 4 weeks.
* People who have ever had radiation treatments to their chest.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People scheduled for endoscopy at Johns Hopkins who have esophageal cancer, Barrett's esophagus or gastro-esophageal reflux disease
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2002-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
early predictors of esophageal cancer | 3
  To see if changes in certain areas of DNA can predict risk for esophageal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Canto, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States